CLINICAL TRIAL: NCT05137392
Title: Impact of Intensive Oral Hygiene Regimen Based on Individualized Messages and an Intelligent Power-driven Toothbrush on Non-surgical Treatment of Stage II and III Periodontitis: A Randomized, Standard of Care-controlled Trial
Brief Title: Effect of Novel Oral Hygiene Regimen on Non-surgical Treatment of Stage II and III Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Maurizio Tonetti, Professor, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: iBrush0817
Record Dates: First submitted 2021-11-03; First posted 2021-11-30 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Periodontitis
Keywords: mobile health; oral hygiene instruction; internet of things network; artificial intelligence
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test group (Experimental): The test group will receive the novel regimen of oral hygiene instruction, including use of a commercially available intelligent toothbrush connected to the Chinese consumer version of an application and receiving targeted oral health message as well as use of interdental toothbrush
  Interventions: Other: oral hygiene instruction
- Control group (Other): The test group will receive the standard regimen of oral hygiene instruction, including use of a commercially available manual toothbrush and receiving a brochure for oral hygiene instruction as well as use of interdental toothbrush
  Interventions: Other: oral hygiene instruction

INTERVENTIONS:
Other: oral hygiene instruction — The treatment process is identical for both test and control groups except for the methods of oral hygiene instructions. In the control group, the participants will receive the following oral hygiene instructions at completion of debridement, at week-1 and week-3. In the test group, apart from the standard oral hygiene instructions at completion of debridement, at week-1 and week-3 , additional analysis of brushing data and provision of targeted brief interventions will be provided on a daily basis for the first week, 3 times/week until week 6 and once a week thereafter until 6 months after the debridement.

SUMMARY:
Achievement of adequate oral hygiene standards is critical to the successful treatment of gum disease. The improvement of the patient's adherence to good oral hygiene is of great importance to obtain the satisfactory treatment outcomes. However, patients' adherence to a proper daily oral hygiene regimen generally remains poor. New electric artificial intelligence powered toothbrushes are able to precisely sense the location of the brushing being performed by the patient and transmit information to the clinician who is able to analyze the data and provide targeted instructions, if needed. This study evaluates whether a novel oral hygiene instruction regimen can provide some additional benefit for periodontal treatment compared with routine oral hygiene instructions.

DETAILED DESCRIPTION:
Dental plaque is causally linked to gingival inflammation and essential for the onset of periodontitis. The main goal of periodontal treatment is the establishment of adequate infection control to reduce the bacterial load below individual threshold levels of inflammation. Achievement of adequate oral hygiene standards is critical to effective periodontal therapy. Classical studies have shown that professional tooth cleaning during healing of subgingival debridement provides superior outcomes. Regrettably, costs do not allow routine implementation of these regimens. By far, patient-centred homecare is the most cost-effective approach to maintaining good oral hygiene. Therefore, improving the adherence with self-performed oral hygiene is a priority in periodontal practice.

Conventionally, clinicians provide oral hygiene instructions to the patients based on the results of their clinical examinations, sometimes supplemented with written information in brochure and disclosing agents to show the location of the biofilm. However, patients' adherence to a proper daily oral hygiene regimen generally remains poor. New technology based on an internet of things network of intelligent toothbrushes (i-Brush) has shown excellent adherence of use in a pilot study in a maintenance population. Other studies have shown that electronic messaging and mobile health (mHealth) supported by smartphones and applications improve oral hygiene performance, particularly in younger individuals undergoing orthodontic treatment. New electric artificial intelligence powered toothbrushes are able to precisely sense the location of the brushing being performed by the patient and transmit information to the clinician who is able to analyze the data and provide targeted instructions, if needed. Remote sensing of oral hygiene practices through the connected intelligent powered toothbrush allows more specific and targeted messages, thereby promoting personalized oral health care and eventually improving the healing outcomes of periodontal therapy through a two-way communication between patients and clinicians. This study aims to investigate the clinical efficacy of a novel regimen consisting of a new generation of power-driven internet connected i-Brush and targeted m-Health messages in improving periodontal treatment outcomes in comparison with routine oral hygiene instructions.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 and above
* Generalized Stage II and Stage III periodontitis
* Subjects willing to receive NSPT necessary for the management of periodontitis and to comply with research appointments/schedule
* Use of a compatible Android cell phone with Oral-B 8.5.1 Application

Exclusion Criteria:

* Edentulism
* Presence of any systemic disease that can alter the manifestation/outcome of periodontal treatment
* Pregnancy or intention to become pregnant at any point during the study duration
* Having received antibiotics within the previous 3 months
* Need for antibiotic prophylaxis in the context of dental treatment
* Having received professional periodontal treatment (other than supragingival cleaning) within the previous 12 months
* Presence of xerostomia interfering with saliva sampling
* Participation in another intervention trial
* Inability or unwillingness of individual to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-10-15 (Actual)

PRIMARY OUTCOMES:
changes in probing pocket depth (PPD) | from baseline to 6 months
  changes in probing pocket depth (PPD) after non-surgical periodontal treatment (NSPT)
changes in proportion of periodontal pocket closure | from baseline to 6 months
  changes in proportion of periodontal pocket closure defined by probing pocket depth (PPD) ≤4mm without bleeding on probing (BOP) after non-surgical periodontal treatment (NSPT)

SECONDARY OUTCOMES:
changes in clinical attachment level (CAL) | from baseline to 6 months
  changes of clinical attachment level (CAL) after non-surgical periodontal treatment (NSPT)
changes in bleeding on probing (BOP) | from baseline to 6 months
  changes in bleeding on probing (BOP) after non-surgical periodontal treatment (NSPT)
changes in periodontal soft tissue volumes | from baseline to 6 months
  changes in periodontal soft tissue volumes or reduction of tissue edema after non-surgical periodontal treatment (NSPT)
changes in oral biomarker concentration | from baseline to 6 months
  the changes in biomarker concentration in saliva and oral rinse after non-surgical periodontal treatment (NSPT)
changes in proportion of periodontal pocket closure | from baseline to 3 months
  changes in proportion of periodontal pocket closure is defined by probing pocket depth (PPD) ≤4mm without bleeding on probing (BOP) after non-surgical periodontal treatment (NSPT)
changes in probing pocket depth (PPD) | from baseline to 3 months
  changes in probing pocket depth (PPD) after non-surgical periodontal treatment (NSPT)

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Tonetti, DMD PhD, Principal Investigator — Shanghai Clinical Research Unit
Locations (1):
- Shanghai PerioImplant Innovation Center, Ninth People Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Toniazzo MP, Nodari D, Muniz FWMG, Weidlich P. Effect of mHealth in improving oral hygiene: A systematic review with meta-analysis. J Clin Periodontol. 2019 Mar;46(3):297-309. doi: 10.1111/jcpe.13083. PMID 30761580
- [Result] Johansson LA, Oster B, Hamp SE. Evaluation of cause-related periodontal therapy and compliance with maintenance care recommendations. J Clin Periodontol. 1984 Nov;11(10):689-99. doi: 10.1111/j.1600-051x.1984.tb01317.x. PMID 6594355
- [Result] Suvan J, Leira Y, Moreno Sancho FM, Graziani F, Derks J, Tomasi C. Subgingival instrumentation for treatment of periodontitis. A systematic review. J Clin Periodontol. 2020 Jul;47 Suppl 22:155-175. doi: 10.1111/jcpe.13245. PMID 31889320
- [Result] Tonetti MS, Deng K, Christiansen A, Bogetti K, Nicora C, Thurnay S, Cortellini P. Self-reported bleeding on brushing as a predictor of bleeding on probing: Early observations from the deployment of an internet of things network of intelligent power-driven toothbrushes in a supportive periodontal care population. J Clin Periodontol. 2020 Oct;47(10):1219-1226. doi: 10.1111/jcpe.13351. Epub 2020 Aug 31. PMID 32748486
- [Result] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- [Result] Sanz M, Herrera D, Kebschull M, Chapple I, Jepsen S, Beglundh T, Sculean A, Tonetti MS; EFP Workshop Participants and Methodological Consultants. Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. J Clin Periodontol. 2020 Jul;47 Suppl 22(Suppl 22):4-60. doi: 10.1111/jcpe.13290. PMID 32383274
- [Derived] Li Y, Wu X, Liu M, Deng K, Tullini A, Zhang X, Shi J, Lai H, Tonetti MS. Enhanced control of periodontitis by an artificial intelligence-enabled multimodal-sensing toothbrush and targeted mHealth micromessages: A randomized trial. J Clin Periodontol. 2024 Dec;51(12):1632-1643. doi: 10.1111/jcpe.13987. Epub 2024 Apr 17. PMID 38631679